CLINICAL TRIAL: NCT00173043
Title: The Role of Insulin Resistance and Adiponectin in the Pathogenesis of Polycystic Ovary Syndrome
Brief Title: The Role of Insulin Resistance in PCOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701208; NSC 94-2314-B-002-195-
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-11-24 (Estimated); Status verified 2004-10

CONDITIONS: Polycystic Ovary Syndrome; Insulin Resistance; Obesity
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Polycystic ovary syndrome (PCOS) phenotype can be structured into three components: anovulation, hyperandrogenism and the metabolic syndrome (of which hyperinsulinemia, secondary to insulin resistance, is the central abnormality)(1). It is the most common endocrinologic disease seen in Gynecologic clinic. The follicular excess in polycystic ovaries and the failure of selection of one dominant follicle contribute to the anovulation of PCOS. The infertile PCOS female usually suffered from difficult ovulation induction and high risk of ovarian hyperstimulation syndrome because of extensive stimulation.

PCOS is the main androgen disorder in women and has been suggested to be associated with a high risk of developing cardiovascular disease and type-2 diabetes. In many PCOS patients, overweight or central obesity is generally associated with increases in fasting insulin levels, insulin resistance, and glucose intolerance, and has been identified as a target for new therapeutic strategy, including early change in lifestyle.

Insulin resistance, defined as decreased insulin-mediated glucose utilization, is commonly (10-25%) found in the normal population. In women with PCOS, insulin resistance appears even more common (up to 50%), in both obese and non-obese women.Hyperinsulinemia appears to play a key pathogenic role in the ovarian androgen overproduction, because of the stimulatory effect of insulin on ovarian steroid production.

DETAILED DESCRIPTION:
Because of the menstrual irregularity and the hirsutism/acne caused by hyperandrogenism, the treatment of choice for PCOS in young teenagers is to given the oral contraceptive; however, such oral contraceptives fail to correct the endocrinometabolic anomalies and the excess of fat. Therefore, there are some alternative treatments as adding the novel progesterone, which is claimed to have antimineralocorticoid and antiandrogenic activities, or giving an insulin-sensitizing compound such as metformin. These treatments were reported to be effective in changing the endocrinometabolic state and the adiposity of PCOS. Besides, they were also reported to have efficacy in aiding ovulation induction.

PCOS is the main androgen disorder in women and has been suggested to be associated with a high risk of developing cardiovascular disease and type-2 diabetes. In many PCOS patients, overweight or central obesity is generally associated with increases in fasting insulin levels, insulin resistance, and glucose intolerance, and has been identified as a target for new therapeutic strategy, including early change in lifestyle.

The plasma concentrations of adiponectin were lower in men than in women but were not different between pre- and postmenopausal women. It suggests that androgen act to reduce plasma adiponectin concentration. In animal experiment, testosterone supplement reduced plasma adiponectin concentration in male mice. In cultured 3T3-L1 adipocytes, testosterone and 5α-DHT suppressed the secretion of adiponectin, suggesting that androgen decreased plasma adiponectin concentration through its effect on adipocytes.

Clinical and/or biochemical signs of hyperandrogenism are one of the three diagnostic criteria defining the PCOS. Hyperandrogenemia may cause hirsutism, alopecia, acne, and also strongly affect the ovulatory function. Some hormone therapy such as ethinylestradiol cyproterone and ethinlyestradiol drosipirenone were usually used to reduce the serum androgen level and correct the amenorrhea/oligomenorrhea, while its effect in improving the endocrine-metabolic state and the adiposity of PCOS was still undetermined. Obese women with PCOS are known to have high serum concentrations of C-reactive protein (CRP), a marker of inflammation and cardiovascular risk factor; metformin monotherapy reduces the CRP levels, whereas combined treatment with ethinylestradiol and cyproterone-acetate raises CRP further. Therefore, I am interesting about how do the metformin and ethinylestradiol/cyproterone acetate influence the serum adiponectin level.

Insulin resistance, defined as decreased insulin-mediated glucose utilization, is commonly (10-25%) found in the normal population. In women with PCOS, insulin resistance appears even more common (up to 50%), in both obese and non-obese women. Criteria developed for defining a metabolic syndrome in PCOS includes components associated with insulin resistance syndrome including centripetal obesity, hypertension, fasting hyperglycemia and dyslipidemia. Since serum adiponectin concentrations correlate inversely with the severity of insulin resistance was well established, however, the adiponectin levels in women with PCOS is still controversial and need further elucidation. Such as Orio et al. suggested that insulin sensitivity does not play any pivotal role in the control of adiponectin in PCOS women and Ducluzeau et al. mentioned that glucose-to-insulin level is better than adiponectin in predicting insulin resistance in PCOS. Besides, adiponectin level reduced in obese women with PCOS was reported. Currently only a clinical trial suggested that the oral contraceptives plus metformin may reduce the adipocytokine imbalance.

Hyperinsulinemia appears to play a key pathogenic role in the ovarian androgen overproduction, because of the stimulatory effect of insulin on ovarian steroid production. The mechanism that allows the ovary to remain sensitive to insulin when classical target organs for insulin action (liver, fat, and muscle) exhibit insulin resistance was supported by the presence of phosphatidyl inositol 3 (PI-3) kinase independent insulin signaling pathway in human ovarian cells (theca and granulosa cell). Insulin is proposed to directly stimulate activity of cytochrome P450c17α, an enzyme involved in ovarian androgen synthesis that is found in thecal cells.

ELIGIBILITY:
Inclusion Criteria:

* Criteria for the definition of PCOS: (2 out of 3 in the following) Oligomenorrhea / chronic anovulation, defined as less than eight cycles of spontaneous menstrual period in one year.

Clinical and /or biochemical signs of hyperandrogenism Polycystic ovaries Exclusion of other aetiologies, such as congenital adrenal hyperplasia, androgen-secreting tumors, Cushing's syndrome

Exclusion Criteria:

* ever received hormone therapy in the past 6 months, having pregnancy in the past 6 months, having acute illness found in the past 3 months, or having systemic diseases including autoimmune disease, malignancy, hepatic, renal or CVS disease, and ever received chemotherapy or immunosuppressive agents.

Ages: 12 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 500
Dates: Start 2004-10; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yu-Shih, M.D., PhD, Principal Investigator — Department of Obstetrics and Gynecology, NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan